CLINICAL TRIAL: NCT01413399
Title: A Pilot Study of Intra-arrest Therapeutic Hypothermia in Patients Suffering Non-Traumatic Out of Hospital Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MeckHypo2011
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2021-11

CONDITIONS: Out-of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-Arrest Therapeutic Hypothermia (Active Comparator)
  Interventions: Drug: 4 degree chilled saline
- Post-Arrest Therapeutic Hypothermia (Active Comparator)
  Interventions: Drug: 4 degree chilled saline

INTERVENTIONS:
Drug: 4 degree chilled saline — 4 degree chilled saline up to 2L in the prehospital setting

SUMMARY:
The objective of this study will be to assess the frequency of return of spontaneous circulation (ROSC), survival to admission, survival to discharge from the hospital, and neurologic function at time of discharge from the hospital among patients experiencing out of hospital cardiac arrest randomized to receive either intra-arrest induction of therapeutic hypothermia (IATH) or post-arrest therapeutic hypothermia (TH).

DETAILED DESCRIPTION:
Therapeutic hypothermia improves mortality and functional neurologic outcomes in patients resuscitated from pulseless ventricular tachycardia and fibrillation (VT/VF), with several studies validating the safety of prehospital induction following successful (return of spontaneous circulation) ROSC by the rapid infusion of 2 liters of 4ºC intravenous fluids. However, the optimal timing for inducing hypothermia remains uncertain. Early studies demonstrated the efficacy of therapeutic hypothermia despite delays of 4 to 8 hours from the time of ROSC to the initiation of cooling. The post-resuscitation reperfusion injury evolves quickly and was thought to be best attenuated by hypothermia induction immediately following return of spontaneous circulation (ROSC). This was supported by animal data which demonstrated that improved neurologic outcome was associated with reduced time to goal temperature following ROSC. More recently this hypothesis has been called into question by 2 clinical trials which suggested that time to initiation of cooling was not associated with improved neurologic outcome at discharge.

There may be another benefit to early therapeutic cooling. Animal data suggest that intra-arrest induction of therapeutic hypothermia (IATH) improves rates of ROSC from cardiac arrest. This is corroborated by a report describing an impressively high ROSC rate of 60.9% among patients receiving IATH. This was a higher frequency of ROSC than reported in similar patient groups. It has been demonstrated that mild hypothermia exerts a stabilizing effect on the myocardium, decreasing the rate of refibrillation following ROSC. Mild hypothermia has also been shown to prolong ventricular refractoriness and repolarization, possibly facilitating electrical defibrillation by slowing repolarization ion currents.

Recently we conducted a retrospective observational study that demonstrated an association between the administration of IATH and ROSC.22 We found that the likelihood of ROSC with IATH was 2.4 (95% CI 1.41-4.24) time higher in the subset of patients who received > 700ml of 4º C normal saline compared to those who did not receive IATH. Our study lacked sufficient power to demonstrate a difference in survival to admission or discharge; however, we noted trends towards improved survival. Current intra-arrest treatments do not obtain ROSC rates greater than those seen in our study with IATH. These associations were noted in all rhythms, including asystole and pulseless electrical activity.

Obtaining ROSC quickly with the resulting decrease in time spent in a low or no flow circulation would have obvious downstream effects on both hospital mortality and neurologic function, independent of the effect of mild hypothermia in the post-arrest inflammatory state. Surprisingly these associations were seen even with fluid volumes that were too low to change core body temperature suggesting that the benefits of therapeutic hypothermia on the myocardium may be possible even at relatively low fluid volumes.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest of presumed medical etiology in the out-of-hospital setting

Exclusion Criteria:

* Traumatic Cardiac Arrests
* Cardiac Arrests Due to hemorrhage
* Cardiac arrests involving children or young adults
* Patients presumed to be pregnant
* Patients with a do not resuscitate

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Studnek, PhD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center; Center for Prehospital MEdicine, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Garrett JS, Studnek JR, Blackwell T, Vandeventer S, Pearson DA, Heffner AC, Reades R. The association between intra-arrest therapeutic hypothermia and return of spontaneous circulation among individuals experiencing out of hospital cardiac arrest. Resuscitation. 2011 Jan;82(1):21-5. doi: 10.1016/j.resuscitation.2010.09.473. Epub 2010 Oct 30. PMID 21036449

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-Arrest Therapeutic Hypothermia: 4 degree chilled saline: 4 degree chilled saline up to 2L in the hospital setting
Period: Overall Study
Arm/Group | Intra-Arrest Therapeutic Hypothermia | Post-Arrest Therapeutic Hypothermia
Started | 208 | 334
Completed | 208 | 334
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra-Arrest Therapeutic Hypothermia | Post-Arrest Therapeutic Hypothermia | Total
Number analyzed (Participants) | 208 | 334 | 542
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 65.9 [63.6 to 68.2] | 63.9 [62.0 to 65.7] | 64.5 [63.0 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 127 | 212
  Male | 123 | 207 | 330
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 208 | 334 | 542

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survived Up To Hospital Discharge
Description: Adjusted OR and 95% CI
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-Arrest Therapeutic Hypothermia | Post-Arrest Therapeutic Hypothermia
Number analyzed (Participants) | 208 | 334
Participants | 24 | 40

2. Secondary Outcome: Number of Patients Who Achieve Prehospital Return of Spontaneous Circulation
Description: ROSC will be defined as return of sustained pulses during the prehospital cardiac arrest resuscitation
Time Frame: Patients will be followed for the duration of their prehospital course of care expected to be an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-Arrest Therapeutic Hypothermia | Post-Arrest Therapeutic Hypothermia
Number analyzed (Participants) | 208 | 334
Participants | 76 | 90

ADVERSE EVENTS:
Arm/Group | Intra-Arrest Therapeutic Hypothermia | Post-Arrest Therapeutic Hypothermia
Serious Adverse Events (participants affected / at risk) | 0/208 | 0/334
Other Adverse Events (participants affected / at risk) | 0/208 | 0/334

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No